CLINICAL TRIAL: NCT06989476
Title: Using Process Mapping to Optimize the Integration of Child Psychosocial Screenings in Primary Care, Promote Whole-person Care, and Increase Family Linkages to Behavioral and Safety Net Services
Brief Title: Process Mapping to Optimize Child Psychosocial Screenings in Primary Care, and Increase Family Service Linkages
Acronym: CARELOOP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Denver Health and Hospital Authority (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-1929; 1R01HS029858-01A1 (AHRQ)
Record Dates: First submitted 2025-04-30; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-04

CONDITIONS: Mental Health Care
Keywords: mental health; pyschosocial needs; service linkage; service mapping; primary care
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: a parallel-arm cluster randomized trial to test the effectiveness of the CARELOOP intervention. Study clinics (11 clusters) will be randomly assigned: 5 clinics will screen children ages 0-5 years and activate referrals per standard care (Control group), and 6 clinics will use Standard Care plus the CARELOOP intervention (Intervention group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CARELOOP Intervention Group (Experimental): Clinics using the CARELOOP intervention to screen children ages 0 to 5 and link children and their caregivers to support services
  Interventions: Other: CARELOOP Intervention
- Standard Care (No Intervention): Clinics screening children ages 0-5 years to identify psychosocial and activate referrals per standard care

INTERVENTIONS:
Other: CARELOOP Intervention — CARELOOP Intervention (Clinics cAtch needs, REfer, Link to services, and close the lOOp using an equitable family-centered Process).
  CARELOOP is a way of enhancing psychosocial screenings through PSM methodology and Implementation Science, and grounded in the Clinical-Community Relationships Evaluation framework
  Arms: CARELOOP Intervention Group

SUMMARY:
Many families screened in primary care for social challenges to identify psychosocial needs of caregivers and children do not receive the follow-up support they need. This study will test a new clinic-based approach, CARELOOP, designed to improve how families are referred to and connected with services. Using community input and a method called Process Service Mapping, the project will tailor clinic workflows and evaluate the approach's impact through a randomized trial. The goal is to improve care coordination and reduce health disparities.

DETAILED DESCRIPTION:
Despite an increased health systems investment in primary care screenings to identify the psychosocial needs of caregivers and children (e.g., exposure to violence, racism, and insecure housing), these efforts don't always result in family-centered service referrals and follow-up to ensure all needs are getting met (i.e., families able to access services such as housing and behavioral health support). When psychosocial needs aren't identified or addressed during childhood, it can cause or worsen children's health conditions, interrupt their development, and, at the societal level, perpetuate disparities in overall health. The investigators' preliminary data identified key strengths and weaknesses within families' journeys through psychosocial screenings, service referral and linkage processes in primary care - which the investigators term "service pathways". The goal of the current study is to optimize the post-screening pathway to increase family referral and linkage follow-up, so that all screened families receive consistent services. The investigators hypothesis is that clinics using the proposed adaptive intervention package will increase family referral and linkage follow-up compared to clinics using current screening practices. A novel and replicable approach to optimize service pathways that include these family-centered elements and implementation strategies is Process Service Mapping (PSM). PSM is an iterative approach to mapping patients' pathways to identify inequities, challenges, and action points. This study seeks to scale up previous work by testing the CARELOOP Intervention (Clinics cAtch needs, REfer, Link to services, and close the lOOp using an equitable family-centered Process). CARELOOP is a system-level intervention that will tailor primary care workflows with PSM-informed decision rules, procedural steps, and implementation strategies with input from clinics and communities. Denver Health is an optimal partner as they are a large safety net system serving minoritized families and 11 pediatric clinics already screen for psychosocial needs using the Health-Related Social Needs and Survey of Well-being of Young Children. The investigators' main hypothesis is that intervention clinics will have higher Service Referrals and Linkages compared to standard care control clinics. After optimizing service pathways (Aim 1), the investigators will conduct a cluster-randomized trial to test the impact of CARELOOP on effectiveness (Aim 2) and implementation outcomes (Aim 3). The study goals are: Aim 1: Engage clinics and communities to refine the CARELOOP intervention by mapping service pathways to include equity and family-centered elements and tailored strategies; Aim 2: Use a parallel-arm cluster randomized trial to test the effectiveness of the CARELOOP intervention; and Aim 3: Conduct an implementation evaluation of the CARELOOP intervention. This R01 study leverages current psychosocial screening practices to rigorously test an intervention designed to increase service referrals and linkages. The investigators bring quality improvement, implementation science, and a novel co-creation engagement approach to accelerate family-centered care

ELIGIBILITY:
Inclusion Criteria:

* Caregiver of child is 18 years or older with legal custody or authority to arrange care for child ages 0-5 years old.
* Caregiver provides informed consent
* Caregiver provides permission for socio-demographic information about their child to be pulled from EMR records, de-identified, and shared with PI

Exclusion criteria

* Caregiver declines to provide signed informed consent, HIPAA release, or permission for socio-demographic data to be pulled from the Electronic Medical Records (EMR), de-identified and shared with PI;
* Children ages 6-18 scheduled for wellness visits
* Children ages 0-5 scheduled for wellness visits outside the study data collection windows or at clinics not providing pediatric care
* Caregiver does not have legal guardianship or written authority to arrange care for the child

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2026-02-17 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Service referral | Through study data collection completion, an average of 2 years; years two through four of the project.
  Number of service referrals / Total number of positive screenings (i.e., caregiver reported a need and accepts outreach for a service referral by clinic navigator).
Service linkage | Through study data collection completion, an average of 2 years; years two through four of the project.
  Caregiver made contact with the referred service

SECONDARY OUTCOMES:
Referral-to-linkage time | Through study data collection completion, an average of 2 years; years two through four of the project.
  Number of days and based on date of referral after screenings (EHR data at the clinic) and date of referral reported by partner Community Based Organizations

CONTACTS AND LOCATIONS:
Locations (1):
- Denver Health, Denver, Colorado, United States